CLINICAL TRIAL: NCT00358475
Title: Study of Perennial Allergic Rhinitis -Long Term Treatment Study-
Brief Title: Study Of Perennial Allergic Rhinitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FFR100688
Record Dates: First submitted 2006-07-27; First posted 2006-07-31 (Estimated); Last update posted 2018-08-31 (Actual); Status verified 2018-08

CONDITIONS: Rhinitis, Allergic, Seasonal
Keywords: perennial allergic rhinitis
MeSH Terms: conditions — Rhinitis, Allergic, Seasonal; Rhinitis, Allergic, Perennial

INTERVENTIONS:
Drug: GW685698

SUMMARY:
This study was designed to assess safety of an investigational nasal spray in the treatment of perennial allergic rhinitis. Perennial allergic rhinitis is triggered by house dust, mite and mold etc. Typical symptoms are sneezing, nasal congestion and pruritus and rhinorrhea.

ELIGIBILITY:
Inclusion criteria:

* Informed consent.
* Outpatient.
* Diagnosis of perennial allergic rhinitis with symptoms.
* Able to comply with study procedures.

Exclusion criteria:

* Significant concomitant medical condition.
* Use of corticosteroids/allergy medications.
* Laboratory abnormality.
* Positive pregnancy test.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2005-06-21; Primary Completion 2005-10-01 (Actual); Study Completion 2005-10-12 (Actual)

PRIMARY OUTCOMES:
Adverse events and laboratory blood test

SECONDARY OUTCOMES:
Change of nasal symptom score

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site